CLINICAL TRIAL: NCT05425875
Title: A Randomized Controlled Trial to Compare Procedural Yield of Bronchoalveolar Lavage Using Three Different Techniques in Subjects Undergoing Flexible Bronchoscopy
Brief Title: Comparison of Procedural Yield of Bronchoalveolar Lavage Using Three Different Techniques in Subjects Undergoing Flexible Bronchoscopy
Acronym: BAL-3T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Inderpaul singh, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: INT/IEC/2021/SPI-1048
Record Dates: First submitted 2022-06-10; First posted 2022-06-21 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Bronchoalveolar Lavaage; Diffuse Lung Disease

STUDY DESIGN:
Intervention Model Description: Three arm parallel group study
Who Masked: Investigator
Masking Description: Investigator will be blinded to the group allotment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manual suction (Experimental): A 50-mL syringe will be used to apply the suction.
  Interventions: Procedure: Bronchoalveolar lavage using manual suction
- Manual suction with tubing (Experimental): A 50-mL syringe with a 15-cm rubber tubing.
  Interventions: Procedure: Bronchoalveolar lavage using manual suction with rubber tubing
- Wall mount suction (Active Comparator): A negative pressure of <100 mmHg will be applied using continuous wall suction.
  Interventions: Procedure: Bronchoalveolar lavage using wall mount suction

INTERVENTIONS:
Procedure: Bronchoalveolar lavage using wall mount suction — BAL will be performed using wall mount suction with a pressure <100 mmHg
  Arms: Wall mount suction
Procedure: Bronchoalveolar lavage using manual suction — A 50-mL syringe will be used to apply suction through the working channel of a bronchoscope
  Arms: Manual suction
Procedure: Bronchoalveolar lavage using manual suction with rubber tubing — A 50-mL syringe with an attached rubber tubing will be used to apply suction through the working channel of a bronchoscope
  Arms: Manual suction with tubing

SUMMARY:
Bronchoalveolar lavage (BAL) via flexible bronchoscopy is a method used to sample the cellular and microbiological components of the alveolar space. It is a procedure in which 2-3 measured aliquots of sterile normal saline are instilled after wedging the scope to the suitable segmental bronchus. BAL is performed from the segments/ lobes showing ground-glass opacities (GGO), tree-in-bud lesions or focal consolidations guided by HRCT. In diffuse lung involvement, BAL is performed either from RML or the lingula.[3] It is recovered through the bronchoscope via different suction methods so as to get a sample of epithelial lining fluid of small airways and alveoli. Either manual suction or wall suction can be used for aspiration of fluid during BAL. The fluid recovered is then sent for cytology and microbiology examination studies including AFB, MGIT, GeneXpert, Galactomannan, fungal cultures to diagnose various conditions like PAP, eosinophilic pneumonia, bacterial or fungal infections, specific forms of ILD.

Three techniques have been described to perform BAL. To the best of our knowledge no previous study has compared the three methods of obtaining the BAL in the same cohort of subjects.The authors believe that the procedural yield of BAL will be best by manual suction using rubber tubing compared to manual suction without rubber tubing or wall suction. Herein, the investigators compare the three methods of obtaining BAL in subjects undergoing BAL for various respiratory diseases

DETAILED DESCRIPTION:
Bronchoalveolar lavage (BAL) via flexible bronchoscopy is a method used to sample the cellular and microbiological components of the alveolar space. It is a procedure in which 2-3 measured aliquots of sterile normal saline are instilled after wedging the scope to the suitable segmental bronchus. BAL is performed from the segments/ lobes showing ground-glass opacities (GGO), tree-in-bud lesions or focal consolidations guided by HRCT. In diffuse lung involvement, BAL is performed either from RML or the lingula.[3] It is recovered through the bronchoscope via different suction methods so as to get a sample of epithelial lining fluid of small airways and alveoli. Either manual suction or wall suction can be used for aspiration of fluid during BAL. The fluid recovered is then sent for cytology and microbiology examination studies including AFB, MGIT, GeneXpert, Galactomannan, fungal cultures to diagnose various conditions like PAP, eosinophilic pneumonia, bacterial or fungal infections, specific forms of ILD Normal BAL cellular components are specified as: Alveolar macrophages (AM) 85%, Lymphocytes 5-15%, Neutrophils <= 3%, eosinophils <1%. The presence of squamous epithelial cells indicates contamination by oropharyngeal secretions. [4] Additionally, BAL can be a tool for pulmonary toilet in rare diseases such as pulmonary alveolar proteinosis by helping to remove the abnormal surfactant material that accumulates with this disease.

Manual suction: It can be done using the same syringe used for instillation of the normal saline. At least 100 ml normal saline should be instilled while performing BAL and should not exceed 200 ml.

According to the studies, Modification of the manual suctioning technique (by connecting small tubing attached to syringe) provides higher percentage of BAL fluid [5].

Wall suction: During suctioning the instilled fluid, negative pressure is applied using continuous wall suction. The pressure should be <100mmHg or should be adjusted to prevent airway collapse.[6] In a study conducted by Aruna D. Herath[7], 73 pediatric patients were enrolled for a RCT undergoing flexible bronchoscopy and BAL. Two different suctioning techniques were compared for % of BAL fluid recovery. Sterile normal saline according to 1ml/kg was instilled and 100-150mmHg of negative pressure was applied for wall suction method. Thus it concluded that wall suction had better BAL fluid recovery than handheld syringe suction. Diagnostic yield was the same for both techniques.

Luis M. Seijo[8], conducted a prospective randomized study of total 220 patients undergoing BAL. Study comparing manual and wall suction in performance of BAL resulted that manual aspiration is superior to wall suction yielding larger quantity of BAL. Additionally, extra tubing with 50 ml syringe was added in manual suction technique and 50mmHg negative pressure was used in wall suction method.

A prospective clinical study of 66 patients by Naghmeh Radhakrishna[9], comparing techniques for optimal BAL performance used 100ml NS (with 4 aliquots) resulted in no significant difference between both techniques.

Another study to compare two aspiration techniques of BAL in children was conducted by Christian Rosas-Salazar[10] on approximately 540 procedures. Their results suggested that handheld syringe suction provide higher % of fluid return when compared to continuous wall suction.

K.S Woods[11], did a randomized, blinded prospective clinical trial on 18 dogs comparing manual and suction pump aspiration techniques for BAL. 35 ml syringe was used to instill 2ml/kg volumes per site for manual aspiration. Negative pressure of maximum 50mmHg was applied for SPA. Thus, concluded the study showing higher % of BALF return by SPA than manual suction with or without tubing. There was no significant difference in diagnostic yield.

One more multicenter randomized study by Antoni Rosell[12] was conducted to recover BAL fluid comparing only syringe and syringe with attached plastic tube (40cm), for more fluid return. Thus, it resulted in 8% more fluid recovery, more yield and less complications with syringe with tubing suction technique.

To the best of author's knowledge no previous study has compared the three methods of obtaining the BAL in the same cohort of subjects. The investigators believe that the procedural yield of BAL will be best by manual suction using rubber tubing compared to manual suction without rubber tubing or wall suction. Herein, the investigators compare the three methods of obtaining BAL in subjects undergoing BAL for various respiratory diseases.

Study question: Is the procedural yield of BAL different between manual suction using rubber tubing compared to manual suction without rubber tubing or wall suction?

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing BAL procedure for various indications using flexible bronchoscopy

Exclusion Criteria:

* Hemodynamic instability (SBP <90mmHg , Baseline Sp02 <92% on room air)
* Failure to provide informed consent
* Platelet count <20,000 per mm3
* Pregnancy
* Subjects already enrolled in any other study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 942 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
To compare proportional procedures in which we obtain optimal yield | 1 hour (during bronchsocopy)
  optimal yield will be defined if there is at least 30% return of volume instilled and adequate sample (<5% bronchial cells)

SECONDARY OUTCOMES:
Diagnostic yield of BAL | 1 month
  Proportion of BAL in each arm that provide a specific diagnosis
Percentage and volume of BAL fluid | 1 hour (during bronchsocopy)
  Percentage of instilled volume of saline for performing BAL that returns while doing BAL and the exact volume of BAL
Proportion of subjects experiencing complications in each arm | 1 month after the procedure
  Complications will include hypoxemia, fever, escalation of care (need for hospitalization, icu admission or airway intubation), airway bleeding, death, and others

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Bronchoscopy suite, PGIMER, Chandigarh
  - Bronchoscopy suite, Chandigarh

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing